CLINICAL TRIAL: NCT00440440
Title: Effect of Androgel on Total and Regional Adipose Tissue and Lean Body Mass in Type 2 Diabetic Patients With Hypogonadism
Brief Title: Effect of Testosterone Gel Replacement on Fat Mass in Males With Low Testosterone Levels and Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study merged with another study
Sponsor: Diabetes Center of the Southwest (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: sandeep dhindsa, Department of Endocrinology and Metabolism
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR-940
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Hypogonadism; Diabetes
Keywords: hypogonadism; diabetes; visceral fat; hepatic fat; lean mass
MeSH Terms: conditions — Hypogonadism; Diabetes Mellitus | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): testosterone gel
  Interventions: Drug: Testosterone gel
- 2 (Placebo Comparator): placebo gel
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Testosterone gel — Testosterone gel to be applied daily, starting does 5g.
  Other Names: Androgel
  Arms: 1
Drug: placebo — placebo gel apply daily
  Arms: 2

SUMMARY:
The purpose of the study is to find out the effect of replacing testosterone in the form of a gel (Androgel®) on the amount of fat mass in males with low testosterone and diabetes.

DETAILED DESCRIPTION:
Hypogonadism is associated with increase in fat mass, decrease in muscle mass, accelerated bone loss, decreased libido and effects on mood. Androgen replacement in this context is clearly beneficial, and numerous studies have demonstrated improvements in bone and muscle mass, reductions in body fat and improvement in insulin sensitivity, libido and mood following treatment. Testosterone replacement leads to a dose-dependent decrease in adipose tissue and increase in muscle mass and strength. The principal focus of the proposed research is to evaluate the effect of androgel on lean body mass and regional adipose tissue mass (including hepatic and visceral fat) in type 2 diabetic patients with hypogonadism, a population that is likely to benefit from a reduction in adipose tissue and an increase in muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* Males with age 35-75 years inclusive.
* Evidence of hypogonadism: Hypogonadism will be defined as low total testosterone (<300 ng/dL) and low calculated free testosterone (below 6.5ng/dL; calculated using testosterone and SHBG). Testosterone levels will be measured between 8 and 10 am. Subjects who have normal total but low free testosterone levels (or vice versa) will be asked to come again after one week to have their testosterone levels re-measured. They will be included in the study in their free and total testosterone levels are low on re-measurement.
* Type 2 diabetes
* Hemoglobin A1c <8.0 %
* Subjects on medications for diabetes will be allowed as long as they are on stable doses of these compounds for at least 6 weeks. The dose of thiazolidinediones will have to be stable for 3 months prior to the study. The dosage of diabetic medications will not be changed during the study.

Exclusion Criteria:

* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks
* Hepatic disease (transaminase > 3 times normal)
* Renal impairment (serum creatinine > 1.5)
* Chronic steroid therapy
* Use of testosterone or other androgens (such as DHEA) in the last 3 months
* Panhypopituitarism
* HIV or hepatitis C
* Subjects will be excluded from the study for history of prostate or breast cancer, gonadal endocrine disorders
* Current or recent history of major psychiatric illness, significant uncontrolled systemic illness
* Sleep apnea
* History of alcoholism or substance abuse within the past year
* History of taking other drugs that might interfere with the results of the study (ie, Lupron, finasteride, spironolactone, cimetidine, antiandrogens, estrogens, p450 enzyme inducers, barbiturates)
* Abnormal prostate evidenced by prostatic symptoms, prostatic masses or induration on rectal examination, elevated levels of prostate specific antigen (>4 ng/mL; subjects with PSA levels between 2.5-4 ng/mL will be permitted if prostate biopsy is negative) or positive biopsy, a urine flow rate of less than 12 mL/s, or an International Prostate Symptom Score greater than 19
* Hematocrit greater than 50%
* Body weight >300 lbs (this is the maximum weight that can be accommodated on DEXA or MRI machines.
* The subject has systolic blood pressure >170mmHg or diastolic blood pressure >100 mmHg while on or off anti-hypertensive treatment.
* Generalized skin disease that could affect the absorption of testosterone gel (ie, psoriasis);
* Morning prolactin level greater than 40 mg/mL
* Subjects with serum fasting triglyceride concentration > 500 mg/dL at screening or with history of hypertriglyceridemia-induced pancreatitis.
* Participation in any other concurrent clinical trial
* Any other life-threatening, non-cardiac disease
* Use of an investigational agent or therapeutic regimen within 30 days or 5 half-lives (which ever is longer) preceding the first dose of study medication.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Mean absolute change in visceral adipose tissue mass in type 2 diabetic subjects with hypogonadism after 6 months of androgel therapy. | 6 months

SECONDARY OUTCOMES:
Study the effect in type 2 diabetic subjects with hypogonadism after 6 months of androgel therapy on: | 6 months
Mean absolute change in hepatic fat measured by NMR spectroscopy. | 6 months
Mean absolute change in total and regional adipose tissue mass measured by DEXA | 6 months
Mean absolute change in total and regional lean body mass measured by DEXA. | 6 months
Mean absolute change in total body and regional (arm, leg, ribs) BMC and BMD | 6 months
Mean absolute change in hip BMC and BMD (mean of two hips) | 6 months
Mean absolute change in spine BMC and lumbar spine (L1-L4) BMD | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhindsa, MBBS, Principal Investigator — Diabetes Center of the Southwest
Locations (1):
- Diabetes Center of the Southwest, Midland, Texas, United States